CLINICAL TRIAL: NCT07200570
Title: Evaluation of a Vaccine Chatbot on HPV Vaccine Confidence and Hesitancy: a Randomized Controlled Trial and Implementation Science Study
Brief Title: Evaluation of a Vaccine Chatbot on HPV Vaccine Confidence and Hesitancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Zhiyuan Hou, Associate Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Fudan-HPV LLM chatbot
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: HPV Vaccine
Keywords: HPV; vaccine confidence; chatbot; randomised controlled trial; implementation science

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Intervention Group (Experimental): Participants in this arm will be granted access to an interactive, LLM-powered HPV vaccine chatbot for a period of three months. They are invited to use the chatbot to ask any questions related to HPV and HPV vaccine to receive personalized and accurate information. The chatbot invitation will be sent every weeks to reinforce the intervention within the first month.
  Interventions: Behavioral: LLM-Powered HPV Vaccine Chatbot
- Control Group (No Intervention): Participants assigned to the control arm will receive standard care but will not have access to the HPV vaccine chatbot during the study period. For ethical considerations, participants in this arm will be offered access to the chatbot after the end of the study.

INTERVENTIONS:
Behavioral: LLM-Powered HPV Vaccine Chatbot — A vaccine chatbot delivered via WeChat or a web browser, designed to provide information and health education about the HPV vaccine. The chatbot is powered by large language models and is trained on an expert-validated knowledge base derived from authoritative sources such as the WHO and China CDC to ensure accuracy. The knowledge base is validated by experts. The chatbot engages users in interactive, conversational dialogue to answer questions and address concerns regarding HPV and HPV vaccines.
  Arms: Chatbot Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if a chatbot powered by artificial intelligence works to improve HPV vaccination among females aged 15 to 26 in China. A randomized controlled trial and implementation science study will be conducted targeting females as participants. The main questions it aims to answer are:

1. Does the vaccine chatbot influence women's confidence, literacy, hesitancy, and uptake of the HPV vaccine.
2. What are the public acceptance of chatbot and the facilitators and barriers to its implementation in a real-world setting.

Researchers will compare a group of women who use the chatbot with a group who do not use it to see if the chatbot is effective at helping women feel confident and willing to get vaccinated against HPV.

Participants will:

1. Be recruited and randomly allocated into one of two groups. One group will be invited to use the HPV vaccine chatbot and the other group will not get access to the vaccine chatbot until the end of the trial.
2. Complete a questionnaire survey on their confidence, literacy, and hesitancy on the HPV vaccine.
3. Have their vaccination status checked at the end of trial.

DETAILED DESCRIPTION:
A randomized controlled trial with 2 arms will be conducted to evaluate the effectiveness of an LLM-powered chatbot on improving HPV vaccination among females aged 15 to 26, followed by a pragmatic implementation science study to assess the public acceptance of chatbot and to identify the facilitators and barriers to its implementation in a real-world setting.

The sample size is calculated based on the primary outcome of the HPV vaccination uptake among females aged 15 to 26 in China. This uptake is around 10% according to the China CDC estimation, and we assume that it can increase to 15% following the intervention. With a significance level (α) of 0.05 and 80% power (1-β=0.8), a sample size of at least 683 per group is needed to detect a 5% absolute difference in vaccination rate (from an assumed baseline rate of 10% to 15% post-intervention). The sample size is inflated to 900 per group to account for potential loss to follow-up and to ensure adequate power for a multi-center design.

Participant recruitment will be conducted across three representative regions of China. For those aged 15 to 18, their parents will be also enrolled. A randomization method will be employed to ensure balanced allocation across two groups, and the randomization sequence will be generated by an independent statistician to ensure a 1:1 allocation ratio.

Participants in the intervention group will be invited to use the HPV vaccine chatbot. The chatbot powered by a large language model (LLM), offers a scalable, accessible, and interactive platform around the HPV vaccine information. The control group will not get access to the vaccine chatbot until the end of the trial. Following the intervention, all participants will complete a questionnaire survey on their confidence, literacy, and hesitancy on the HPV vaccine. And their vaccination status will be obtained from official vaccination records at the end of trial.

The intention-to-treat (ITT) analysis will be used to evaluate the effectiveness of the intervention. Between-group comparisons will use t-tests for continuous variables and chi-square tests for categorical variables. To adjust for potential confounders, generalized estimating equation (GEE) models will be employed to provide robust effect estimates. Timing of vaccination will be evaluated using Kaplan-Meier survival curves and log-rank tests, with Cox proportional hazards models to estimate intervention effects on time-to-vaccination. Subgroup analyses will assess heterogeneity of intervention effects across populations stratified by baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 15 to 26 years, inclusive.
* Not previously vaccinated against HPV.
* Reports no contraindications to HPV vaccination.
* Has no mental, visual, or reading impairments that would preclude cooperation with study activities.
* Is willing and able to provide informed consent.

Exclusion Criteria:

* Male.
* Age under 15 or over 26 years.
* Has a history of prior HPV vaccination.
* Has a known contraindication to HPV vaccination.
* Unable to comply with study procedures.
* Is unwilling or unable to provide informed consent.

Ages: 15 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HPV Vaccine Uptake | Three months after participant randomization allocation
  Whether participants get vaccinated against HPV, measured by official vaccination records.

SECONDARY OUTCOMES:
HPV Vaccine Hesitancy | The same day after the intervention
  HPV vaccine hesitancy will be measured using a 5-point Likert scale that assesses a participant's willingness to receive the HPV vaccine, with options ranging from "very willing" to "very unwilling". A higher score on the scale indicates higher hesitancy.
HPV Vaccine Confidence | The same day after the intervention
  Vaccine Confidence Index (VCI) that assesses confidence in the importance, effectiveness, and safety of vaccines using a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A higher score indicates greater confidence.
HPV Vaccine Literacy | The same day after the intervention
  A series of questions about HPV vaccine knowledge and misinformation. Total literacy score is calculated based on the number of questions answered correctly by the participants.
Timing of HPV Vaccination | Within three months after participant randomization allocation
  When participants get vaccinated against HPV, measured by official vaccination records
Chatbot Usability | The same day after the intervention
  A series of questions assessing usability and feasibility, fairness and safety, user experience, and overall assessment of the chatbot.
Cost of interventions | Within three months after participant randomization allocation
  The cost of designing and implementing chatbot interventions. Unit of Measure: Chinese Yuan (CNY).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant privacy concerns and institutional data protection policies.

REFERENCES:
- [Background] Weeks R, Sangha P, Cooper L, Sedoc J, White S, Gretz S, Toledo A, Lahav D, Hartner AM, Martin NM, Lee JH, Slonim N, Bar-Zeev N. Usability and Credibility of a COVID-19 Vaccine Chatbot for Young Adults and Health Workers in the United States: Formative Mixed Methods Study. JMIR Hum Factors. 2023 Jan 30;10:e40533. doi: 10.2196/40533. PMID 36409300
- [Background] Weeks R, Cooper L, Sangha P, Sedoc J, White S, Toledo A, Gretz S, Lahav D, Martin N, Michel A, Lee JH, Slonim N, Bar-Zeev N. Chatbot-Delivered COVID-19 Vaccine Communication Message Preferences of Young Adults and Public Health Workers in Urban American Communities: Qualitative Study. J Med Internet Res. 2022 Jul 6;24(7):e38418. doi: 10.2196/38418. PMID 35737898
- [Background] Kobayashi T, Nishina Y, Tomoi H, Harada K, Tanaka K, Matsumoto E, Horimukai K, Ishihara J, Sasaki S, Inaba K, Seguchi K, Takahashi H, Salinas JL, Yamada Y. Corowa-kun: A messenger app chatbot delivers COVID-19 vaccine information, Japan 2021. Vaccine. 2022 Jul 30;40(32):4654-4662. doi: 10.1016/j.vaccine.2022.06.007. Epub 2022 Jun 8. PMID 35750541
- [Background] Almalki M, Azeez F. Health Chatbots for Fighting COVID-19: a Scoping Review. Acta Inform Med. 2020 Dec;28(4):241-247. doi: 10.5455/aim.2020.28.241-247. PMID 33627924
- [Background] Wilson L, Marasoiu M. The Development and Use of Chatbots in Public Health: Scoping Review. JMIR Hum Factors. 2022 Oct 5;9(4):e35882. doi: 10.2196/35882. PMID 36197708
- [Background] Luk TT, Lui JHT, Wang MP. Efficacy, Usability, and Acceptability of a Chatbot for Promoting COVID-19 Vaccination in Unvaccinated or Booster-Hesitant Young Adults: Pre-Post Pilot Study. J Med Internet Res. 2022 Oct 4;24(10):e39063. doi: 10.2196/39063. PMID 36179132
- [Background] Si M, Su X, Jiang Y, Wang W, Zhang X, Gu X, Ma L, Li J, Zhang S, Ren Z, Liu Y, Qiao Y. An Internet-Based Education Program for Human Papillomavirus Vaccination Among Female College Students in Mainland China: Application of the Information-Motivation-Behavioral Skills Model in a Cluster Randomized Trial. J Med Internet Res. 2022 Sep 30;24(9):e37848. doi: 10.2196/37848. PMID 36178723
- [Background] Si M, Su X, Jiang Y, Wang W, Zhang X, Gu X, Ma L, Li J, Zhang S, Ren Z, Liu Y, Qiao Y. Effect of an IMB Model-Based Education on the Acceptability of HPV Vaccination Among College Girls in Mainland China: A Cluster RCT. Cancer Control. 2022 Jan-Dec;29:10732748211070719. doi: 10.1177/10732748211070719. PMID 35088609
- [Background] Wang D, Wu J, Du J, Ong H, Tang B, Dozier M, Weller D, Campbell C. Acceptability of and barriers to human papillomavirus vaccination in China: A systematic review of the Chinese and English scientific literature. Eur J Cancer Care (Engl). 2022 May;31(3):e13566. doi: 10.1111/ecc.13566. Epub 2022 Mar 1. PMID 35229931
- [Background] Zhang X, Liu CR, Wang ZZ, Ren ZF, Feng XX, Ma W, Gao XH, Zhang R, Brown MD, Qiao YL, Geng Q, Li J. Effect of a school-based educational intervention on HPV and HPV vaccine knowledge and willingness to be vaccinated among Chinese adolescents : a multi-center intervention follow-up study. Vaccine. 2020 Apr 29;38(20):3665-3670. doi: 10.1016/j.vaccine.2020.03.032. Epub 2020 Mar 31. PMID 32245644
- [Background] Zhang X, Wang Z, Ren Z, Li Z, Ma W, Gao X, Zhang R, Qiao Y, Li J. HPV vaccine acceptability and willingness-related factors among Chinese adolescents: a nation-wide study. Hum Vaccin Immunother. 2021 Apr 3;17(4):1025-1032. doi: 10.1080/21645515.2020.1812314. Epub 2020 Oct 29. PMID 33121330
- [Background] Wei Z, Liu Y, Zhang L, Sun X, Jiang Q, Li Z, Wu Y, Fu C. Stages of HPV Vaccine Hesitancy Among Guardians of Female Secondary School Students in China. J Adolesc Health. 2023 Jan;72(1):73-79. doi: 10.1016/j.jadohealth.2022.08.027. Epub 2022 Oct 11. PMID 36229401
- [Background] Xie Y, Su LY, Wang F, Tang HY, Yang QG, Liu YJ. Awareness regarding and vaccines acceptability of human papillomavirus among parents of middle school students in Zunyi, Southwest China. Hum Vaccin Immunother. 2021 Nov 2;17(11):4406-4411. doi: 10.1080/21645515.2021.1951931. Epub 2021 Jul 29. PMID 34324411
- [Background] Zhang Y, Wang Y, Liu L, Fan Y, Liu Z, Wang Y, Nie S. Awareness and knowledge about human papillomavirus vaccination and its acceptance in China: a meta-analysis of 58 observational studies. BMC Public Health. 2016 Mar 3;16:216. doi: 10.1186/s12889-016-2873-8. PMID 26936076
- [Background] Zang S, Zhang X, Qu Z, Chen X, Hou Z. Promote COVID-19 Vaccination for Older Adults in China. China CDC Wkly. 2022 Sep 16;4(37):832-834. doi: 10.46234/ccdcw2022.173. No abstract available. PMID 36284538
- [Background] Sonawane K, Zhu Y, Montealegre JR, Lairson DR, Bauer C, McGee LU, Giuliano AR, Deshmukh AA. Parental intent to initiate and complete the human papillomavirus vaccine series in the USA: a nationwide, cross-sectional survey. Lancet Public Health. 2020 Sep;5(9):e484-e492. doi: 10.1016/S2468-2667(20)30139-0. Epub 2020 Jul 21. PMID 32707126
- [Background] Drolet M, Benard E, Perez N, Brisson M; HPV Vaccination Impact Study Group. Population-level impact and herd effects following the introduction of human papillomavirus vaccination programmes: updated systematic review and meta-analysis. Lancet. 2019 Aug 10;394(10197):497-509. doi: 10.1016/S0140-6736(19)30298-3. Epub 2019 Jun 26. PMID 31255301
- [Background] Falcaro M, Castanon A, Ndlela B, Checchi M, Soldan K, Lopez-Bernal J, Elliss-Brookes L, Sasieni P. The effects of the national HPV vaccination programme in England, UK, on cervical cancer and grade 3 cervical intraepithelial neoplasia incidence: a register-based observational study. Lancet. 2021 Dec 4;398(10316):2084-2092. doi: 10.1016/S0140-6736(21)02178-4. Epub 2021 Nov 3. PMID 34741816
- [Background] Chen Y, Jiang N, Jiao Y, Chen J, Cao A, An J, Dang Y. Analysis of HPV vaccination and influencing factors among 9-14-year-old girls in underdeveloped areas of northwestern China: A cross-sectional survey report on guardians. Vaccine. 2025 Aug 30;62:127568. doi: 10.1016/j.vaccine.2025.127568. Epub 2025 Aug 7. PMID 40780093
- [Background] Hu S, Xu X, Zhang Y, Liu Y, Yang C, Wang Y, Wang Y, Yu Y, Hong Y, Zhang X, Bian R, Cao X, Xu L, Zhao F. A nationwide post-marketing survey of knowledge, attitude and practice toward human papillomavirus vaccine in general population: Implications for vaccine roll-out in mainland China. Vaccine. 2021 Jan 3;39(1):35-44. doi: 10.1016/j.vaccine.2020.11.029. Epub 2020 Nov 23. PMID 33243631